CLINICAL TRIAL: NCT01764100
Title: Mesenchymal Stromal Cells (MSC) for the Treatment of Severe (Grade II-IV) Steroid-resistant Graft Versus Host Disease (GVHD): a Phase I Trial
Brief Title: Mesenchymal Stromal Cells (MSCs) for the Treatment of Graft Versus Host Disease (GVHD)
Acronym: MSC-GvHD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ettore Biagi, MD (Other)
Responsible Party: Sponsor-Investigator, Ettore Biagi, MD, Ettore Biagi, MD, Azienda Ospedaliera San Gerardo di Monza
Organization: Azienda Ospedaliera San Gerardo di Monza (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-MSC; 2008-007869-23 (EudraCT Number)
Record Dates: First submitted 2010-05-05; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal Stromal Cells (MSC) (Experimental): Intravenous injections for a dose of 1 ± 0.5 x 106 MSC/kg recipient body weight
  Interventions: Genetic: Mesenchymal stromal cells

INTERVENTIONS:
Genetic: Mesenchymal stromal cells — Mesenchymal stromal cells (MSC) intravenous infusion at least two fixed doses of mesenchymal stem cells (1 ± 0.5 x 106/kg recipient body weight for each injection) with 5 to 7 days of interval one from the other, derived from HLA unrelated donor different from the HSC donor (third party donor).

SUMMARY:
This is a bicentric, prospective, non randomized study. Pediatric and adult patients will be treated.

Rationale: MSC have shown promising effects by reversal of severe therapy-resistant acute GvHD. As a common therapeutic line of action is not shared for steroid resistant GVHD, it is important to establish the toxicity and the feasibility of preparation and infusion of third party MSCs for acute steroid resistant GVHD and acute phases of chronic steroid resistant GVHD.

A total of 10 patients (pediatric and adults) need to be enrolled in the study. Patients who present clinical signs of either acute or chronic steroid resistant GVHD will receive by intravenous infusion at least two fixed doses of mesenchymal stem cells with 5 to 7 days of interval one from the other, derived from HLA unrelated donor different from the HSC donor (third party donor) regardless of the rate of HLA mismatch.

Primary objectives are to establish the feasibility and the toxicity of preparation and infusions of third party MSCs for the treatment of steroid resistant acute and acute phases of chronic grade II-IV GVHD.

Secondary objectives are:

1. To document the efficacy of MSC infusion in steroid resistant acute and acute phases of chronic GVHD grade II-IV.
2. To document the rate of GVHD recurrence in MSCs infused patients.
3. To document relapse of hematological malignancies post MSC infusions in patients undergoing MSCs treatment for steroid refractory GvHD.
4. To document the overall survival of MSC infused patients for steroid refractory GvHD.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Patients are required to meet the following inclusion criteria:

Any patient that has undergone allogeneic stem cell transplantation with steroid refractory grades II-IV acute GvHD either occurring post transplant, or induced by donor lymphocyte infusions (DLI) or T-cell add back, or chronic steroid refractory GVHD in acute phase. Patients may be receiving local best treatment for steroid refractory GVHD. A positive biopsy for GvHD is not required if clinical signs and symptoms are characteristic for GvHD and other etiologies are excluded. See 6.4 for acute GvHD grading.

1. Steroids have been given, for instance methylprednisolone 2 mg/kg/day, for at least 72h in case of progressive acute GvHD, 5 days in case of stable acute GVHD (grade II to IV) or chronic GvHD in active phase, according to the local policy.
2. Despite this treatment, the patient has unresponsive GvHD after 5 days, or progressive acute GvHD after 72 hours. If single organ acute GvHD grade II from gut or liver, either progression from single organ or addition of one or two more organs. As an example, if the patient has grade II acute GvHD of the skin, GvHD is more intense and more widespread, or GvHD also includes liver and/or gut.
3. Patients with steroid refractory GvHD fulfilling the requirements mentioned in a) - b) may be treated with second line therapy according to the clinical guidelines at each center prior to enrolment in this study.
4. Patients under treatment with best available local treatment for steroid resistant GVHD will not interrupt the ongoing treatment unless clinically required for safety reasons.

Exclusion Criteria:

1. Inability to obtain informed consent.
2. Patients with documented uncontrolled EBV, CMV or fungal infection.
3. Patients in poor clinical conditions with life expectancy of less than 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Any toxic effect reported during MSCs infusion or in the subsequent 10 days by clinical monitoring | During MSCs infusion or in the subsequent 10 days
Feasibility as the possibility of producing adequate lots of patient dedicated MSCs for any patients presenting with steroid resistant GVHD | three years

SECONDARY OUTCOMES:
Number of patients with GvHD resolution | One month
  1. Complete resolution of GvHD: Control of all signs and symptoms attributed to acute GvHD
  2. Partial resolution of GvHD: Control of some signs and symptoms attributed to acute GvHD with an improvement of overall grade
  3. Refractory GvHD: No change in signs or symptoms of GvHD within 10 days of MSC infusion.
  4. Worsening GvHD: Any progress of GvHD signs and symptoms that increase overall grade. a and b will be defined as response. c and d will be defined as no response.
Determination of recurrence of GvHD | After 1 month from MSCs infusion
Relapse of haematological disease | Every three months
Survival | Every three months

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Biagi, MD, Principal Investigator — San Gerardo Hospital
Locations (3):
- Italy (3):
  - U.O. Ematologia - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Clinica Pediatrica CTMO - Azienda Ospedaliera San Gerardo, Monza, MB
  - U.O. Ematologia CTMO - Azienda Ospedaliera San Gerardo, Monza, MB

REFERENCES:
- [Derived] Introna M, Lucchini G, Dander E, Galimberti S, Rovelli A, Balduzzi A, Longoni D, Pavan F, Masciocchi F, Algarotti A, Mico C, Grassi A, Deola S, Cavattoni I, Gaipa G, Belotti D, Perseghin P, Parma M, Pogliani E, Golay J, Pedrini O, Capelli C, Cortelazzo S, D'Amico G, Biondi A, Rambaldi A, Biagi E. Treatment of graft versus host disease with mesenchymal stromal cells: a phase I study on 40 adult and pediatric patients. Biol Blood Marrow Transplant. 2014 Mar;20(3):375-81. doi: 10.1016/j.bbmt.2013.11.033. Epub 2013 Dec 7. PMID 24321746